CLINICAL TRIAL: NCT06854991
Title: Neuroimaging Biomarkers for Assessing Brain Mechanisms Mediating Virtual Reality Anxiety and Pain Management
Brief Title: Healthy Children and Virtual Reality Mediation of Simulated Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Henry Xiang, Director, Center for Pediatric Trauma Research, Nationwide Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00004727
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Pain; Experimental Pain in Healthy Human Participants; Children; Adolescents
Keywords: Acute Pain; Experimental Pain; Virtual Reality; fNIRS
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: All participants will start with a control condition (no distraction tool) and will then receive an Active VR, Passive VR, and iPad game distraction in random order during their experimental pain/fNIRS session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will wear an fNIRS neuroimaging device and undergo an experimental pain session using a blood pressure cuff around the calf. No distraction tool will be used.
- Active VR-PAT (Experimental): Participants will wear an fNIRS neuroimaging device and undergo an experimental pain session using a blood pressure cuff around the calf. Participants actively play an engaging virtual reality game on a VR headset.
  Interventions: Other: Active VR-PAT
- Passive VR-PAT (Active Comparator): Participants will wear an fNIRS neuroimaging device and undergo an experimental pain session using a blood pressure cuff around the calf. Participants view a video of the same VR game on a VR headset, without engagement.
  Interventions: Other: Passive VR-PAT
- iPad game (Active Comparator): Participants will wear an fNIRS neuroimaging device and undergo an experimental pain session using a blood pressure cuff around the calf. Participants actively play the same VR game on an iPad, without the immersion of a VR headset.
  Interventions: Other: iPad

INTERVENTIONS:
Other: Active VR-PAT — Virtual Reality Pain Alleviation Tool (VR-PAT) hosted on a Pico Neo 3 Pro Eye headset. Both engagement and immersion.
  Arms: Active VR-PAT
Other: Passive VR-PAT — VR-PAT hosted on a Pico Neo 3 Pro Eye headset, with the active game participation removed. Immersion with engagement removed.
  Arms: Passive VR-PAT
Other: iPad — VR-PAT hosted on an Apple iPad. Engagement with immersion removed.
  Arms: iPad game

SUMMARY:
The objective of this study is to develop central nervous system (CNS) biomarkers of pain experienced during medical procedures and pain relief induced by Virtual Reality Pain Alleviation Therapy (VR-PAT). The study team plans to use innovative functional near-infrared spectroscopy (fNIRS) to identify and quantify the targeted CNS biomarkers. The ultimate goal of this project is to optimize the CNS biomarkers for predicting and/or monitoring response to virtual reality (VR)-based pain reduction approaches for pain management in clinical trials.

20 healthy children will be recruited for a 1-hour research visit where they will wear a blood pressure cuff to simulate pain and an fNIRS neuroimaging device while playing an immersive/engaging VR game, a passive VR video, and an iPad game.

DETAILED DESCRIPTION:
The objective of this study is to develop central nervous system (CNS) biomarkers of pain experienced during medical procedures and pain relief induced by Virtual Reality Pain Alleviation Therapy (VR-PAT). The study team plans to use innovative functional near-infrared spectroscopy (fNIRS) to identify and quantify the targeted CNS biomarkers. The ultimate goal of this project is to optimize the CNS biomarkers for predicting and/or monitoring response to VR-based pain reduction approaches for pain management in clinical trials.

Collaboration will occur through a team science model to address the following three specific aims:

Aim 1: To quantify the central nervous system (CNS) responses associated with self-reported pain intensity during a simulated pain condition.

Aim 2: To assess brain response patterns to virtual reality (VR)-based interventions for pain management.

Aim 3: To assess the degree to which objective brain measures and brain responses to VR intervention modulate objective brain markers of pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years, inclusive
* Subjects and legal guardians can communicate (read and write) using English

Exclusion Criteria:

* Currently experiencing any pain (acute or chronic)
* Took any pain medication within the past 12 hours
* Vision, hearing, or cognitive/motor impairments preventing valid administration of study measures
* History of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
* Minors in foster care, incarcerated, or currently pregnant

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in brain activation picked up on fNIRS between the active VR, passive VR, iPad game, and control conditions | Assessed continuously throughout the simulated pain session (60 minutes) for one visit
  Mean within subject fNIRS signals of brain activation

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, MBA, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No